CLINICAL TRIAL: NCT06333665
Title: Correlation Analysis of Type II Diabetes Mellitus on Short-term and Long-term Outcomes of Patients With Esophageal Squamous Cell Cancer Undergoing Minimally Invasive Esophagectomy
Brief Title: PPIO-007 Correlation Analysis of Type II Diabetes Mellitus on Short-term and Long-term Outcomes of Patients With Esophageal Squamous Cell Cancer Undergoing Minimally Invasive Esophagectomy
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, WEI GUO, chief physician, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: Wei G
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamous Cell Carcinoma; Surgery
Keywords: Esophageal Squamous Cell Carcinoma; diabetes mellitus; surgery; postoperative complications; survival outcomes
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Diabetes Mellitus; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coe-T2DM group: There was a definitive diagnosis of type 2 diabetes mellitus before surgery
  Interventions: Other: Whether there is type 2 diabetes mellitus before surgery
- No-T2DM group: There was no clear diagnosis of type 2 diabetes mellitus before surgery

INTERVENTIONS:
Other: Whether there is type 2 diabetes mellitus before surgery — Patients were grouped according to whether they had type 2 diabetes mellitus before surgery
  Groups: Coe-T2DM group

SUMMARY:
To date, there is controversy as to whether type II diabetes mellitus is associated with adverse short- and long-term outcomes in patients with esophageal squamous cell carcinoma undergoing minimally invasive esophagectomy. At the same time, to the best of our knowledge, the impact of metformin use and glycemic control on short- and long-term outcomes in this patient population is also controversial. Therefore, this study aims to test the hypothesis that diabetes mellitus is associated with reduced survival in patients with esophageal squamous cell carcinoma undergoing minimally invasive esophagectomy and that treatment with metformin and/or good glycemic control (HbA1c<7.0%) is associated with improved survival.

DETAILED DESCRIPTION:
Esophageal cancer is one of the major components of the global cancer burden. According to the Global Cancer Statistics 2020 report, in 2020, esophageal cancer ranked ninth in the world in incidence (604,100 new cases) and sixth in overall mortality (544,076 deaths). In China, esophageal cancer ranked fifth among cancer-related causes of death in 2020, with more than 90% of esophageal cancers being esophageal squamous cell carcinoma (ESCC). Until now, surgery-based comprehensive treatment has remained the main mode of treatment for patients with potentially curable localized esophageal cancer. However, despite efforts to advance treatment, the five-year survival rate for patients with esophageal cancer after surgery is still low, so it is important to identify prognosis-related factors.

Diabetes is a global health problem that has reached alarming levels. In 2019, nearly half a billion people worldwide (9.3% of adults aged 20-79 years) had diabetes, with approximately 20% in the age group aged 60-75 years (the main incidence group of esophageal cancer). Diabetes mellitus is a wasting systemic disease associated with poor outcomes across multiple disease processes and is one of the greatest challenges facing healthcare systems worldwide. For malignant tumors, diabetes is not only one of the causes but also one of the risk factors for low survival. Although other cancer specialties (eg, colon, pancreatic, breast) are associated with poor oncology outcomes, it may be due to decreased immunity and increased systemic inflammation in patients with diabetes. However, there is controversy regarding the prognostic role of diabetes mellitus in patients undergoing surgery for esophageal cancer. There is evidence that patients with diabetes have an increased risk of cancer recurrence and death after surgery compared with non-diabetic controls; However, some studies have shown no significant association between T2DM and postoperative complications, suggesting that diabetes is not an independent risk factor for survival.

Metformin, a member of the biguanide family, is commonly used as an oral antihyperglycemic agent that reduces cancer risk and improves prognosis for a variety of cancers. In recent years, the use of metformin has improved survival in patients with malignant tumors. For patients with esophageal squamous cell carcinoma (ESCC), several molecular mechanisms have been shown to inhibit tumor progression, for example, by inhibiting the growth of esophageal cancer cells. Metformin has also been shown to have a beneficial prognostic effect on some other tumors, such as colon, lung, and prostate cancers, in some studies. The association between metformin use and mortality in patients undergoing surgery for esophageal cancer has been analyzed with conflicting results. A study by Van De Voorde et al. showed that the use of metformin was associated with significantly better distant metastasis-free survival and overall survival. In contrast, the results of Spierings et al. showed that metformin use did not result in higher pathologic response rates or improved overall survival or disease-free survival. They believe that contrary to the assumptions of other tumor types, metformin may not have a beneficial effect on esophageal cancer.

Studies have shown that T2DM does not appear to have a significant effect on the long-term survival of esophageal cancer patients undergoing esophagectomy. In contrast, it may be more important to control blood glucose levels in patients with T2DM undergoing esophagectomy. At the same time, a large number of studies have confirmed that diabetic patients with poor glycemic control have a higher complication rate after esophageal cancer surgery, especially anastomotic leakage.

In summary, there is controversy as to whether type II diabetes mellitus will result in adverse short- and long-term outcomes for patients with esophageal squamous cell carcinoma undergoing minimally invasive esophagectomy. At the same time, to the best of our knowledge, the impact of metformin use and glycemic control on short- and long-term outcomes in this patient population is also controversial. Therefore, this study aims to test the hypothesis that diabetes mellitus is associated with reduced survival in patients with esophageal squamous cell carcinoma undergoing minimally invasive esophagectomy and that treatment with metformin and/or good glycemic control (HbA1c<7.0%) is associated with improved survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clear pathologic diagnosis of esophageal squamous cell carcinoma;
2. Received minimally invasive McKeown procedure;
3. Patients with R0 resection (R0: radical resection).

Exclusion Criteria:

1. Concomitant history of other primary cancers or other cancers;
2. Distant metastases before surgery;
3. Serious comorbidities of other systems before surgery;
4. Patients diagnosed with T2DM during follow-up;
5. The medical record information is incomplete.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EC who attended the Department of Thoracic Surgery at Daping Hospital and underwent the McKeown MIE procedure performed by the same surgical team were included for evaluation from September 2017 to September 2021.
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Overall survival | About five years postoperatively
  Overall survival (OS) was defined as the time from the date of surgery to death from any cause or last follow-up.
Disease-free survival | About five years postoperatively
  Disease-free survival (DFS) was defined as the time from the date of surgery to recurrence, metastasis, and death from any cause.

SECONDARY OUTCOMES:
postoperative adverse events | within 90 days postoperatively
  including pneumonia, adult respiratory distress syndrome (ARDS), anastomotic leak (AL), vocal cord paralysis, chylothorax, pneumothorax, pleural effusion, cardiovascular complications
perioperative 90-day mortality | within 90 days postoperatively
  Mortality within 90 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Army Medical Center of the People's Liberation Army, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No